CLINICAL TRIAL: NCT01831648
Title: An Open, Prospective, National, Multicenter, Non Randomised, Study Based on Healthy Volunteers for Establishing Normative Data for IGF1 in the General Population
Brief Title: Establishment of Reference Values for Insulin-like Growth Factor 1 (IGF1) in the General Population
Acronym: VARIETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: P081216
Record Dates: First submitted 2013-04-03; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Population
Keywords: IGF1; standards; Assays; Z-score; Healthy volunteers; Population
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volonteers (Experimental): Blood sample
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
Various assays can be used for IGF-I measurement in French laboratories. Unfortunately, each assay gives a very different result for the same sample. As IGF-I also varies with age, it is necessary to establish a broad population reference values of IGF1 concentration for each of the IGF1 assays used in clinical practice, taking into account individual variation factors such as age, nutritional status and possible treatments.

The objective of this study is to establish normative data based on a large random selection from the general population, including representation from all age groups (around 100 subjects for each decade age range). This will be performed for all the available assay kits. Subjects with medical conditions and medications that may affect the outcome will be excluded. Normative data will include the range (2.5 to 97.5 percentiles) in mass units and results will be reported as mass units but also as SD scores in order to be able, in a given patient, to compare its IGF-I concentration along time, even if using different assays.

DETAILED DESCRIPTION:
Healthy subjects will be recruited in 30 centers all around France. A total of 1000 healthy subjects are necessary. Each subject will have a clinical examination with measurement of height and weight. Personal medical history will be recorded and gonadal status evaluated. Biological standard workup will be performed and 80 ml of blood will be sampled and serum will be aliquoted, frozen and stored at -80°C. IGF-I level will be measured with all the assay methods available (sera kept in bank will be used in the future when new methods will be available) For each assay method and each age group (Four 3-years groups between 18 and 30 years and six decade age groups between 30 and 89 years) IGF-I will be measured.

Results will be expressed as mean, median, standard deviation, 2.5th and 97.5th percentiles, in mass units. Modelisation according to age and other factors will be performed in order to allow the reporting of IGF-I results for a given individual expression of IGF-I as Z-score.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 89 years old (18 years ≤ age ≤ 89 years)
* Consent given by the patient
* No history of : thyroid disease, liver disease or kidney disease or metabolic endocrine disease cardiovascular or pulmonary disease, neoplastic disease, gastroenterological disease (malabsorption, parasites, chronic diarrhea, peptic disease), psychiatric illness, epilepsy.
* No medication that can interfere with the concentration of IGF1: steroids, anti-androgens, distal diuretics, anti-estrogens, enzyme inducers (rifampin, rifabutin, phenobarbital, phenytoin, carbamazepine, herbal St. John's wort, efavirenz, nevirapine, griseofulvin , OP'DDD, mitotane).
* No intercurrent illness in the week preceding the inclusion
* No known chronic infectious disease (BVH, CVH, HIV)
* No active smoking
* Weight/height2 (BMI) less than 28 kg/m2 and greater than 19 kg/m2
* Normal clinical examination
* Normal blood pressure: children under 65 years (100 mm Hg <SBP <140 mmHg, 50 mmHg <PAD <90 mmHg) for over 65 years (100 mm Hg <SBP <150 mmHg, 50 mmHg <SBP <90mmHg )

Exclusion Criteria:

* Uncontrolled intercurrent illness
* Pregnant or lactating woman
* Excess alcohol consumption: more than 50 g/24h of chronic or acute or unable to restraint from consuming alcohol
* Susceptible to use drugs
* Donated blood in the 3 months preceding the study
* Blood transfusion in the 3 months preceding the test
* Exclusion period of a previous experimental trial.
* Fasting extended by several days.
* Patient not affiliated to a social security system (is or should be beneficiary)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Concentration of IGF1 in serum | up to 4 hours
  Establishment of reference values for the concentration of IGF1 in the general adult population for each of the assays of IGF1 used in clinical practice, taking into account individual variation factors such as age, nutritional status and potential treatments.

SECONDARY OUTCOMES:
Development of an expression results in Z-score for all assays to overcome the differences related to different immunoassays. | up to 4 hours
Establishment of a bank of frozen sera to further develop these standards | up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHANSON, Professor, Principal Investigator — Assistance Publique Hôpitaux de Paris - Bicêtre Hospital
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Sabbah N, Wolf P, Piedvache C, Trabado S, Verdelet T, Cornu C, Souberbielle JC, Chanson P. Reference values for IGF-I serum concentration in an adult population: use of the VARIETE cohort for two new immunoassays. Endocr Connect. 2021 Aug 26;10(9):1027-1034. doi: 10.1530/EC-21-0175. PMID 34343107
- [Derived] Loeb E, Becquemont L, Corruble E. Is the decrease in NOx due to a lack of substrate or a NOS inhibition in patients with major depression? : Commentary on Hess et al. 2017. Psychopharmacology (Berl). 2021 Feb;238(2):613-614. doi: 10.1007/s00213-020-05747-x. Epub 2021 Jan 9. No abstract available. PMID 33420804
- [Derived] Loeb E, El Asmar K, Trabado S, Gressier F, Colle R, Rigal A, Martin S, Verstuyft C, Feve B, Chanson P, Becquemont L, Corruble E. Nitric Oxide Synthase activity in major depressive episodes before and after antidepressant treatment: Results of a large case-control treatment study. Psychol Med. 2022 Jan;52(1):80-89. doi: 10.1017/S0033291720001749. Epub 2020 Jun 11. PMID 32524920
- [Derived] Mariette X, Perrodeau E, Verner C, Struillou X, Picard N, Schaeverbeke T, Constantin A, Ravaud P, Bouchard P. Role of good oral hygiene on clinical evolution of rheumatoid arthritis: a randomized study nested in the ESPOIR cohort. Rheumatology (Oxford). 2020 May 1;59(5):988-996. doi: 10.1093/rheumatology/kez368. PMID 31504982
- [Derived] Mavromati M, Kuhn E, Agostini H, Brailly-Tabard S, Massart C, Piketty ML, Arnoux A, Young J, Souberbielle JC, Chanson P. Classification of Patients With GH Disorders May Vary According to the IGF-I Assay. J Clin Endocrinol Metab. 2017 Aug 1;102(8):2844-2852. doi: 10.1210/jc.2017-00202. PMID 28505364
- [Derived] Chanson P, Arnoux A, Mavromati M, Brailly-Tabard S, Massart C, Young J, Piketty ML, Souberbielle JC; VARIETE Investigators. Reference Values for IGF-I Serum Concentrations: Comparison of Six Immunoassays. J Clin Endocrinol Metab. 2016 Sep;101(9):3450-8. doi: 10.1210/jc.2016-1257. Epub 2016 May 11. PMID 27167056